CLINICAL TRIAL: NCT00208156
Title: An Open-Label Extension Study of the Safety and Tolerability of CORLUX™ (Mifepristone) for Recurrent Psychotic Symptoms in Patients With Major Depressive Disorder With Psychotic Features
Brief Title: A United States Extension Study of Corlux for Recurrent Psychotic Symptoms in Psychotic Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-1073-10
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Major Depression; Psychotic Major Depression; PMD; Psychosis
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Psychotic Disorders | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mifepristone (Experimental)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
Corlux (mifepristone) is a new medication that modulates the body's use of a hormone called cortisol. Under normal conditions, cortisol and other hormones are created by the body in response to physical and emotional stress, triggering a healthy stress response. People who suffer from psychotic major depression may have unusually high levels of cortisol circulating within them or abnormal patterns of cortisol levels, overloading the stress response mechanism and causing symptoms of psychosis such as delusional thoughts or hallucinations. If Corlux can keep the body's cortisol receptors from being overloaded, the stress response system may return to normal function, which may result in improvement of symptoms. The purpose of this study is to allow patients who have already participated in an earlier 8 week study of Corlux versus placebo (an inactive pill) to receive additional courses of treatment with Corlux periodically if a psychotic episode should reappear during a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation through Day 56 in Corcept Therapeutics Protocol C-1073-07
* Are 18 to 75 years of age
* Have a diagnosis of major depressive disorder with psychotic features (DSM-IV 296.24 or 296.34)
* Are able to provide written informed consent

Exclusion Criteria:

* Have a major medical problem
* Have a history of an allergic reaction to Corlux (C-1073, mifepristone)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of Corlux (mifepristone) for the treatment of recurrent psychotic symptoms with major depression with psychotic features (PMD) who previously participated in Corcept Therapeutics Protocol C-1073-07

SECONDARY OUTCOMES:
To assess the frequency of retreatment with Corlux in patients with PMD and qualitatively describe the psychotic symptoms for which retreatment is clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Beebe, PhD, Study Director — Corcept Therapeutics
Locations (13):
- United States (13):
  - Cnri, Llc, San Diego, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Robert Horne M.D., Las Vegas, Nevada
  - CNS Research Institute (CRI), Clementon, New Jersey
  - New Jersey Medical School - UMDNJ, Newark, New Jersey
  - BioBehavioral Health, Toms River, New Jersey
  - Zucker Hillside Hospital, Glen Oaks, New York
  - Neurobehavioral Research, Inc., Lawrence, New York
  - IPS Research Company, Oklahoma City, Oklahoma
  - CNS Research Institute (CRI), Philadelphia, Pennsylvania
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - International Clinical Research Associates, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Background] Belanoff JK, Rothschild AJ, Cassidy F, DeBattista C, Baulieu EE, Schold C, Schatzberg AF. An open label trial of C-1073 (mifepristone) for psychotic major depression. Biol Psychiatry. 2002 Sep 1;52(5):386-92. doi: 10.1016/s0006-3223(02)01432-4. PMID 12242054
- [Background] Brogden RN, Goa KL, Faulds D. Mifepristone. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic potential. Drugs. 1993 Mar;45(3):384-409. doi: 10.2165/00003495-199345030-00007. PMID 7682909
- [Background] Belanoff JK, Flores BH, Kalezhan M, Sund B, Schatzberg AF. Rapid reversal of psychotic depression using mifepristone. J Clin Psychopharmacol. 2001 Oct;21(5):516-21. doi: 10.1097/00004714-200110000-00009. PMID 11593077
- See also: Corcept Therapeutics — http://www.corcept.com